CLINICAL TRIAL: NCT05222867
Title: Angle Labor Pain Questionnaire Turkish Version: Validity and Reliability Study and Evaluation of Efficacy With a Non-pharmacological Method
Brief Title: The Effect of Lower Back Massage on Perceived Labor Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Burcu Tuncer Yilmaz, Principal Investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ALPQT_NONFARMA
Record Dates: First submitted 2021-12-14; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): pregnant women undergoing lower back massage
  Interventions: Procedure: lower back massage
- control group (No Intervention): pregnant women given routine care

INTERVENTIONS:
Procedure: lower back massage — Lower back massage performance: In the study, Linda Kimber's massage protocol was used. First, the researcher ensured that the patient was holding the bed, squatting, or bent over on the bed, which is suitable for the massage, between two contractions. The pregnant woman was instructed to breathe deeply and exhale audibly when her contractions began. Gloves were worn during the massage and liquid Vaseline, which does not contain any active substance, was used to provide lubricity. The circular hip massage was applied at the beginning of the contraction, and lower lateral area and sacral pressure massage was applied towards the end of the contraction as per the massage protocol, and simultaneously with the inhaling sound of the pregnant woman
  Arms: Intervention

SUMMARY:
The aim of the study was to assesment the change in pain scores with lower back massage, a non-pharmacological method, on perceived labor pain in the early active phase of the first stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* The study group consisted of pregnant women who were at 37-40 weeks of pregnancy,
* had cervical dilatation of 4-6 cm,
* had a single, live, and vertex fetus,
* had an uncomplicated pregnancy,
* had no contraction anomalies,
* could communicate in Turkish
* planned for a vaginal delivery.

Exclusion Criteria:

* with cognitive dysfunction
* using narcotic analgesics or sedative drugs
* had any contraindications for applying a back massage

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 60 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
assessment of change in pain scores with lower back massage | Change in perceived labor pain scores in an average of 30 minutes (During the lower back massage application)
  Lower back massage is a non-pharmacological method to reduce perceived labor pain.

CONTACTS AND LOCATIONS:
Overall Officials: NEBAHAT OZERDOGAN, PROF.DR., Study Director — ESKISEHIR OSMANGAZI UNIVERSITY FACULTY OF HEALTH SCIENCES DEPARTMENT OF MIDWIFERY
Locations (1):
- Burcu Tuncer Yilmaz, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angle PJ, Kurtz Landy C, Djordjevic J, Barrett J, Kibbe A, Sriparamananthan S, Lee Y, Hamata L, Zaki P, Kiss A. Performance of the Angle Labor Pain Questionnaire During Initiation of Epidural Analgesia in Early Active Labor. Anesth Analg. 2016 Dec;123(6):1546-1553. doi: 10.1213/ANE.0000000000001679. PMID 27870739
- [Background] Angle P, Landy CK, Charles C, Yee J, Watson J, Kung R, Kronberg J, Halpern S, Lam D, Lie LM, Streiner D. Phase 1 development of an index to measure the quality of neuraxial labour analgesia: exploring the perspectives of childbearing women. Can J Anaesth. 2010 May;57(5):468-78. doi: 10.1007/s12630-010-9289-1. Epub 2010 Mar 13. PMID 20229219
- [Background] Capogna G, Camorcia M, Stirparo S, Valentini G, Garassino A, Farcomeni A. Multidimensional evaluation of pain during early and late labor: a comparison of nulliparous and multiparous women. Int J Obstet Anesth. 2010 Apr;19(2):167-70. doi: 10.1016/j.ijoa.2009.05.013. Epub 2010 Mar 9. PMID 20219349
- [Result] Angle P, Kurtz-Landy C, Djordjevic J, Barrett J, Kibbe A, Sriparamananthan S, Lee Y, Hamata L, Kiss A. The Angle Labor Pain Questionnaire: Reliability, Validity, Sensitivity to Change, and Responsiveness During Early Active Labor Without Pain Relief. Clin J Pain. 2017 Feb;33(2):132-141. doi: 10.1097/AJP.0000000000000386. PMID 27685468

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT05222867/Prot_SAP_000.pdf